CLINICAL TRIAL: NCT05067348
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Clinical Trial of the Efficacy and Safety of Tocilizumab in the Treatment of Generalized Myasthenia Gravis
Brief Title: Efficacy and Safety of Tocilizumab in the Treatment of Generalized Myasthenia Gravis
Acronym: tMG
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: V4.0, 20220410
Record Dates: First submitted 2021-09-23; First posted 2021-10-05 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Myasthenia Gravis, Generalized
Keywords: Generalized Myasthenia Gravis; Tocilizumab
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tocilizumab (Experimental): Participants will receive tocilizumab administered intravenously (IV) on weeks 1,5,9 and 13 of the randomized controlled period.
  Interventions: Drug: Tocilizumab Injectable Product
- Placebo (Placebo Comparator): Participants will receive placebo administered intravenously (IV) on weeks 1,5,9 and 13 of the randomized controlled period.
  Interventions: Drug: Tocilizumab Injectable Product

INTERVENTIONS:
Drug: Tocilizumab Injectable Product — Participants will receive IV tocilizumab

SUMMARY:
Randomized, double-blind, placebo-controlled, parallel-group study with optional open-label extension.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled study, to be conducted at 6 study sites. Approximately 64 subjects will be enrolled. Patients with MG who are positive for anti-AChR antibodies will be enrolled. Patients who do not have anti-AChR or anti-MuSK antibodies will not be enrolled. Patients with MGFA classification II, III, or IV disease, MG-ADL score ≥ 5, QMG score ≥ 11, and use of a corticosteroid and/or non-steroidal immunosuppressant will be included in the study.

All subjects who complete the randomized controlled period will have the option to enroll in a 1-year open-label period.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of MG with anti-AChRantibody.
2. MGFA Clinical Classification Class II, III, or IV.
3. MG-ADL score of 5 or greater at screening and at randomization with > 50% of this score attributed to non-ocular items.
4. QMG score of 11 or greater.
5. Subjects must be on:

   1. Cholinesterase inhibitor, with no dose increase within 4 weeks prior to randomization;
   2. Corticosteroids, with no dose increase within 4 weeks prior to randomization; or/and c. non-steroidal IST (including azathioprine, mycophenolate mofetil, tacrolimus, cyclosporine A), with continuous use for at least 6 months prior to randomization and no dose increase within 4 months prior to randomization.

Exclusion Criteria:

1. Participants had clinically relevant active infections (such as sepsis, pneumonia, or abscess) or severe infections (resulting in hospitalization or requiring antibiotic treatment) in the 4 weeks before randomization;
2. Those with a history of high-risk tuberculosis infection, acquired tuberculosis infection, and chronic hepatitis;
3. Human immunodeficiency virus (HIV) infection;
4. Thymomas that have received thymectomy or planned thymectomy during RCP within 6 months before randomization, or require chemotherapy and/or radiotherapy at any time;
5. Received rituximab treatment in the past 6 months before randomization;
6. Received tocilizumab or eculizumab treatment within 3 months before randomization;
7. Received IVIG or plasma exchange within 4 weeks before randomization;
8. Unresected thymoma.
9. History of other tumor diseases.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-07-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Change in Quantitative Myasthenia Gravis (QMG) scores. | 16 weeks

SECONDARY OUTCOMES:
Proportion of subjects with both (1) ≥ 3-point improvement in QMG and (2) lasts ≥4 weeks | 16 weeks
Proportion of subjects with both (1) ≥ 2-point improvement in MG-ADL and (2) lasts ≥4 weeks | 16 weeks
Change from baseline in Myasthenia Gravis Activities of Daily Living (MG-ADL) Profile score. | 16 weeks
Change in Myasthenia Gravis Composite (MGC) score | 16 weeks
Change in Myasthenia Gravis Quality of Life-15, revised (MGQOL-15r) score. | 16 weeks
Change in Myasthenia Gravis Impairment Index (MGII) score. | 16 weeks
Number of participants with treatment-emergent adverse events (TEAEs), adverse events of special interest (AESIs), and treatment-emergent serious adverse events (TESAEs) during the randomized controlled period and open-label period. | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ting Chang, MD,PHD, Study Director — The Second Affiliated Hospital of Air Force Medical University
Locations (6):
- China (6):
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Tangdu Hospital, The Fourth Military Medical University, Xi'an, Shaanxi
  - Huashan Hospital, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Tianjin medical university general hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No